CLINICAL TRIAL: NCT01181531
Title: A Multicenter, Randomized, Open Label Study to Compare the Efficacy of Cinacalcet Versus Traditional Vitamin D Therapy for Management of Secondary Hyperparathyroidism Among Subjects Undergoing Hemodialysis
Brief Title: Compare the Efficacy of Cinacalcet vs Traditional Vitamin D for Secondary Hyperparathyroidism (SHPT) Among Subjects Undergoing Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20090686; PARADIGM (Other: Amgen)
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Hyperparathyroidism, Secondary
Keywords: Secondary Hyperthyroidism; Hemodialysis; Parathyroid; PARADIGM
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — Cinacalcet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Vitamin D Therapy (Active Comparator)
  Interventions: Drug: Traditional Vitamin D Therapy
- Cinacalcet (Experimental)
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: Traditional Vitamin D Therapy — Traditional vitamin D therapy (eg, calcitriol, paricalcitol, alfacalcidol, doxercalciferol), to manage secondary hyperparathyroidism (SHPT) in this study will be administered according to strategies that have been used in clinical practice and that conform to current therapeutic recommendations and available clinical practice guidelines and product labeling.
  Arms: Traditional Vitamin D Therapy
Drug: Cinacalcet — Subjects randomized to treatment with cinacalcet will receive an initial oral dose of 30 mg once daily. Doses will be titrated incrementally to 60, 90,120, and 180 mg per day based upon periodic measurements of serum calcium and plasma PTH levels. Cinacalcet is formulated as light green tablets in 30, 60, and 90 mg free-based equivalents. Tablets will be 30, 60, and 90 mg, graduated in size, smallest to largest. Combinations of these 3 fixed dosage formulations will be used to achieve the 120 and 180 mg daily doses.
  Arms: Cinacalcet

SUMMARY:
The purpose of this study is to determine the efficacy of treatment with cinacalcet to manage plasma parathyroid levels as to compared traditional vitamin D therapy, whether given orally or intravenously, among hemodialysis subjects with secondary hyperparathyroidism when the doses are adjusted appropriately to maintain serum calcium and phosphorous levels with currently recommended ranges.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at screening
* Treated with maintenance hemodialysis 3 times a week for ≥ 3 months prior to screening
* Informed consent provided by the study candidate
* For subjects NOT receiving cinacalcet and/or vitamin D therapy for SHPT within 60 days prior to enrollment: Plasma PTH levels ≥ 450 pg/mL (50 pmol/L) during screening, as obtained from the central laboratory and, Serum corrected total calcium ≥ 8.4 mg/dL (2.1 mmol/L) and < 10.2 mg/dL (2.55 mmol/L) during screening, as obtained from the central laboratory

Exclusion Criteria:

* Parathyroidectomy in the 12 weeks before the date of informed consent
* History of seizure within 12 weeks prior to randomization
* Scheduled for kidney transplant
* Parathyroidectomy anticipated within the next 6 months
* Liver function tests > than 2 x the Upper Limit of Normal
* Prior use of bisphosphonates, or expected to receive bisphosphonates during the trial
* Subject has previously enrolled in this study
* General
* Other investigational procedures are excluded
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational agent(s)
* Subject (male or female) is not willing to use highly effective contraception during treatment and for at least one month (women) and 3 months (men) after the end of treatment
* Subject is pregnant or breast feeding, or planning to become pregnant during study or within 1 month after the end of treatment Male subject with a pregnant partner who is not willing to use a condom during treatment and for at least 1 month after the end of treatment
* Subject has known sensitivity or intolerance to any of the protocol required therapies
* Subject will not be available for protocol-required study visits, to the best of the subject and investigator's knowledge
* Subject has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2012-07-17 (Actual); Study Completion 2012-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Wetmore JB, Gurevich K, Sprague S, Da Roza G, Buerkert J, Reiner M, Goodman W, Cooper K. A Randomized Trial of Cinacalcet versus Vitamin D Analogs as Monotherapy in Secondary Hyperparathyroidism (PARADIGM). Clin J Am Soc Nephrol. 2015 Jun 5;10(6):1031-40. doi: 10.2215/CJN.07050714. Epub 2015 Apr 22. PMID 25904755
- [Derived] Sprague SM, Wetmore JB, Gurevich K, Da Roza G, Buerkert J, Reiner M, Goodman W, Cooper K. Effect of Cinacalcet and Vitamin D Analogs on Fibroblast Growth Factor-23 during the Treatment of Secondary Hyperparathyroidism. Clin J Am Soc Nephrol. 2015 Jun 5;10(6):1021-30. doi: 10.2215/CJN.03270314. Epub 2015 Apr 14. PMID 25873267
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 08 September 2010 through 14 August 2012 Two participants in each arm did not receive Investigational Product (IP) and Traditional Vitamin D.
Groups:
- Traditional Vitamin D: Vitamin D sterol, intravenous (IV) or oral
- Cinacalcet: Cinacalcet Hydrochloride (Sensipar)
Period: Overall Study
Arm/Group | Traditional Vitamin D | Cinacalcet
Started | 157 (Subjects are randomized after washout.) | 155 (Subjects are randomized after washout.)
Received Investigational Product | 155 | 153
Completed | 96 | 102
Not Completed | 61 | 53
Not completed — Other | 17 | 12
Not completed — Partial consent by subject withdrawn | 0 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Noncompliance | 2 | 2
Not completed — Ineligibility determined | 1 | 2
Not completed — Protocol Specified Criteria | 15 | 8
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Protocol Violation | 6 | 6
Not completed — Death | 9 | 12
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Vitamin D | Cinacalcet | Total
Number analyzed (Participants) | 157 | 155 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] — All Enrolled subjects
  years | 54.3 (13.9) | 53.5 (14.5) | 53.9 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 62 | 124
  Male | 95 | 93 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 32 | 79
  Not Hispanic or Latino | 110 | 123 | 233
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 60 | 76 | 136
  White | 86 | 66 | 152
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Mean PTH During Efficacy Assessment Phase (EAP)
Description: Mean PTH during EAP is defined as the mean of values at study weeks 40, 44, 48 and 52
Time Frame: Baseline to week 40-52
Population: All subjects randomized by treatment arm.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Cinacalcet: Cinacalcet Hydrochloride
Arm/Group | Traditional Vitamin D | Cinacalcet
Number analyzed (Participants) | 157 | 155
Percent change | -7 (4.0) | -12.1 (4.0)
Statistical Analysis 1: Comparison: Traditional Vitamin D vs Cinacalcet; Null hypothesis: no difference in % change from baseline in PTH comparing the two treatment arms; Test type: Superiority or Other; p = 0.346, Mixed Models Analysis — Unadjusted. Model contains baseline stratification factor for type of Vitamin D administered at the site; Mean Difference (Final Values) = -5.0, 95% CI 2-sided [-15.4 to 5.4], Standard Error of Mean 5.3 — Cinacalcet - Vitamin D

2. Secondary Outcome: Treatment Comparison of >=30% Reduction From Baseline in Mean PTH During the Efficacy Assessment Phase (EAP)
Description: Number of participants achieving a >=30% Reduction From Baseline in Mean PTH During Efficacy Assessment Phase (EAP)
Time Frame: Baseline to week 40-52
Measure: Number; unit: Participants
Arm/Group | Traditional Vitamin D | Cinacalcet
Number analyzed (Participants) | 157 | 155
Participants
  Yes | 53 | 66
  No | 104 | 89
Statistical Analysis 1: Comparison: Traditional Vitamin D vs Cinacalcet; Test type: Superiority or Other; p = 0.110, Cochran-Mantel-Haenszel — Stratified by type of Vitamin D at site; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.92 to 2.29] — OR is Cinacalcet: Vitamin D

3. Secondary Outcome: Treatment Comparison of Plasma PTH < 300 pg/mL During Efficacy Assessment Phase (EAP)
Description: Number of participants achieving Plasma PTH < 300 pg/mL During Efficacy Assessment Phase (EAP)
Time Frame: week 40-52
Measure: Number; unit: Participants
Arm/Group | Traditional Vitamin D | Cinacalcet
Number analyzed (Participants) | 157 | 155
Participants
  Yes | 24 | 30
  No | 133 | 125
Statistical Analysis 1: Comparison: Traditional Vitamin D vs Cinacalcet; Test type: Superiority or Other; p = 0.346, Cochran-Mantel-Haenszel — stratified by type of Vitamin D at site; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.74 to 2.39] — OR is Cinacalcet: Vitamin D

ADVERSE EVENTS:
Time Frame: 56 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
  Two participants in each arm did not receive Investigational Product (IP) and Traditional Vitamin D.
Arm/Group | Traditional Vitamin D | Cinacalcet
Serious Adverse Events (participants affected / at risk) | 68/155 | 60/153
Other Adverse Events (participants affected / at risk) | 83/155 | 98/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Traditional Vitamin D (N=155) | Cinacalcet (N=153)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 3
Angina pectoris (Cardiac disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 2
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 2
Cardiac discomfort (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 3
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Nodal arrhythmia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 3
Chills (General disorders) | 0 | 1
Death (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 1 | 4
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Thrombosis in device (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 1
Arteriovenous fistula site infection (Infections and infestations) | 2 | 1
Arteriovenous graft site infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 1
Diabetic gangrene (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 2
Sepsis (Infections and infestations) | 2 | 3
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 2 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 4 | 1
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 2 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 5 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal hernia repair (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypertensive emergency (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 3
Ischaemic limb pain (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Traditional Vitamin D (N=155) | Cinacalcet (N=153)
Anaemia (Blood and lymphatic system disorders) | 5 | 4
Hyperparathyroidism (Endocrine disorders) | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 7 | 8
Diarrhoea (Gastrointestinal disorders) | 16 | 15
Nausea (Gastrointestinal disorders) | 10 | 27
Vomiting (Gastrointestinal disorders) | 5 | 16
Asthenia (General disorders) | 1 | 7
Chest pain (General disorders) | 5 | 6
Oedema (General disorders) | 5 | 2
Oedema peripheral (General disorders) | 5 | 8
Pain (General disorders) | 2 | 6
Pyrexia (General disorders) | 8 | 3
Urinary tract infection (Infections and infestations) | 3 | 5
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 7 | 8
Fall (Injury, poisoning and procedural complications) | 4 | 7
Procedural hypotension (Injury, poisoning and procedural complications) | 7 | 4
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 4 | 6
Decreased appetite (Metabolism and nutrition disorders) | 5 | 3
Fluid overload (Metabolism and nutrition disorders) | 8 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 7 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 6
Hyperphosphataemia (Metabolism and nutrition disorders) | 7 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 10
Dizziness (Nervous system disorders) | 5 | 7
Headache (Nervous system disorders) | 4 | 8
Anxiety (Psychiatric disorders) | 8 | 4
Insomnia (Psychiatric disorders) | 6 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 17
Hypertension (Vascular disorders) | 7 | 8
Hypotension (Vascular disorders) | 6 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.